CLINICAL TRIAL: NCT01626885
Title: A Long-Term Study of MP-214 in Patients With Receiving Multiple Drugs Schizophrenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A002-A8
Record Dates: First submitted 2012-06-19; First posted 2012-06-25 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Antipsychotic Agents; Mental Disorder; Psychotropic Drugs; Dopamine Agents; Central Nervous System Agents
MeSH Terms: conditions — Schizophrenia; Mental Disorders

ARMS (1):
- MP-214 1.5-9 mg (Experimental)
  Interventions: Drug: MP-214

INTERVENTIONS:
Drug: MP-214 — Patients who meet eligibility criteria will be administered a once daily oral fixed dose (3mg) of MP-214 for four weeks, then flexible dose (1.5-9 mg) of MP-214

SUMMARY:
The objective of this study is to evaluate the long-term safety, tolerability, and efficacy of MP-214 in patients with receiving multiple drugs schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient before the initiation of any study-specific procedures
* Patients diagnosed with schizophrenia according to the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia
* Patients who receive 1 or more antipsychotic drugs
* Patients with normal physical examination, laboratory, vital signs, and/or electrocardiogram (ECG)

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of schizoaffective disorder, schizophreniform disorder, other psychotic disorders other than schizophrenia, or bipolar I or II disorder

The information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kurayoshi, Tottori, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MP-214 1.5-9 mg
Started | 42
Completed | 30
Not Completed | 12
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | MP-214 1.5-9 mg
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Time Frame: Up to 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MP-214 1.5-9 mg
Number analyzed (Participants) | 42
Participants | 42

ADVERSE EVENTS:
Arm/Group | MP-214 1.5-9 mg
Serious Adverse Events (participants affected / at risk) | 2/42
Other Adverse Events (participants affected / at risk) | 37/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 1.5-9 mg (N=42)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Schizophrenia (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MP-214 1.5-9 mg (N=42)
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Nasopharyngitis (Infections and infestations) | 18
Contusion (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 6
Gamma-glutamyltransferase increased (Investigations) | 3
Weight increased (Investigations) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Akathisia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 3
Extrapyramidal disorder (Nervous system disorders) | 6
Headache (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 3
Initial insomnia (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 5
Irritability (Psychiatric disorders) | 3
Schizophrenia (Psychiatric disorders) | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other